CLINICAL TRIAL: NCT00800306
Title: Levosimendan and Inhaled Nitric Oxide for Resuscitating the Microcirculation in Septic Shock. A Randomized Controlled Trial
Brief Title: Effects of Levosimendan on Microcirculation in Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Andrea Morelli, University of Rome "La Sapienza"
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1102
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Septic Shock
Keywords: sepsis; septic shock; microcirculation; levosimendan; dobutamine; inotropes; inhaled nitric oxide
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Simendan; Dobutamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- levosimendan (Experimental)
  Interventions: Drug: Levosimendan
- Control (Active Comparator)
  Interventions: Drug: dobutamine

INTERVENTIONS:
Drug: Levosimendan — Intravenous administration of Levosimendan 0,2 µg•kg-1•min-1 for 24 hrs followed by the addition of 35 ppm of inhaled nitric oxide
  Arms: levosimendan
Drug: dobutamine — Intravenous administration of dobutamine 5 µg•kg-1•min-1 for 36 hrs. At the end of the first 24 hrs drug infusion, inhaled nitric oxide at the concentration of 35 ppm will be added for further 12 hrs.
  Arms: Control

SUMMARY:
The present study was conducted as a prospective, randomized, controlled study to:

* investigate the effects of a combination of levosimendan and inhaled nitric oxide on systemic hemodynamics and microcirculation in patients with catecholamine-dependent septic shock;
* test the hypothesis that levosimendan plus inhaled nitric oxide may be effective in restoring microvascular function in septic shock.

DETAILED DESCRIPTION:
40 septic shock patients requiring norepinephrine to maintain mean arterial pressure between 65 and 75 mmHg despite adequate volume resuscitation will be enrolled in the study. After an initial hemodynamic resuscitation aimed at achieve a mean arterial pressure between 65 and 75 mmHg and a mixed venous oxygen saturation (SvO2) ≥ 65%, patients will be randomly allocated to be treated with either a) intravenous administration of levosimendan 0.2 µg∙kg-1∙min-1 for 24 hrs, b)intravenous administration of dobutamine 5 µg∙kg-1∙min-1 for 36 hrs(control; each n = 20). At the end of the first 24 hrs of the study period, both groups will receive inhaled nitric oxide at the concentration of 35 ppm for further 12 hrs. In all patients norepinephrine was titrated to maintain mean arterial pressure between 65 and 75 mmHg. Data from right heart catheterization and sublingual microvascular network will be obtained just before randomization (baseline) and then after 24 and 36 hours.

The sublingual microvascular network will be studied using the sidestream dark field (SDF) imaging. The device will be applied on the lateral side of the tongue, in an area approximately 2-4 cm from the tip of the tongue. Sequences of 10 secs from eight adjacent areas will be recorded on disk using a personal computer. These sequences will be later analyzed by an investigator blinded to the patient's diagnosis and therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Septic shock
* Vasopressor support to maintain mean arterial pressure (MAP) between 65 and 75 mmHg despite adequate volume resuscitation (pulmonary artery occlusion pressure = 13-18 mmHg and central venous pressure = 8-12 mmHg)

Exclusion Criteria:

* Pregnancy
* Age < 18 years
* Ventricular outflow tract obstruction
* Mitral valve systolic anterior motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Systemic hemodynamic and Microcirculatory flow index of small and medium vessels (MFI) | over a period of 36 hrs from the time of randomization

SECONDARY OUTCOMES:
Acid-base homeostasis | over a period of 36 hrs from the time of randomization
Oxygen transport variables | over a period of 36 hrs from the time of randomization
Functional capillary density (mm/mm2) (FCD) | over a period of 36 hrs from the time of randomization
De Backer score | over a period of 36 hrs from the time of randomization
Perfused Vessel Density (PVD) (mm/mm2) | over a period of 36 hrs from the time of randomization
Proportion of Perfused vessels (%) (PPV) | over a period of 36 hrs from the time of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, M.D., Principal Investigator — University of Rome "La Sapienza", Department of Anesthesiology and Intensive Care
Locations (1):
- Departement of Anesthesiology and Intensive Care of the University of Rome "La Sapienza" Viale del Policlinico 155, Rome, Italy

REFERENCES:
- [Derived] Morelli A, Donati A, Ertmer C, Rehberg S, Lange M, Orecchioni A, Cecchini V, Landoni G, Pelaia P, Pietropaoli P, Van Aken H, Teboul JL, Ince C, Westphal M. Levosimendan for resuscitating the microcirculation in patients with septic shock: a randomized controlled study. Crit Care. 2010;14(6):R232. doi: 10.1186/cc9387. Epub 2010 Dec 23. PMID 21182783